CLINICAL TRIAL: NCT02136043
Title: A Randomized Study (With Active Treatment in Both Treatment Groups) to Evaluate How a New Vibration Treatment in the Nose in Patients With Non-allergic Rhinitis Can be Done as Convenient as Possible to the Patient
Brief Title: Kinetic Oscillation Stimulation (KOS) of Nasal Mucosa in Non-allergic Rhinitis: Investigation of Treatment Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halmstad County Hospital (Other)
Responsible Party: Principal Investigator, Finn Jorgensen, Finn Jorgensen, M.D., Ph.D., Halmstad County Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHC14.
Record Dates: First submitted 2014-05-05; First posted 2014-05-12 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Non-allergic Rhinitis.
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Insertion of catheter into nasal cavity carried out by patient. Fixation of catheter during treatment with patient´s hand.
  Interventions: Device: PBASE system 1.1 (active treatment)
- Group 2 (Experimental): Insertion of catheter into nasal cavity carried out by health professional. Fixation of catheter during treatment with helmet.
  Interventions: Device: PBASE system 1.1 (active treatment)

INTERVENTIONS:
Device: PBASE system 1.1 (active treatment)

SUMMARY:
The purpose of the study is to evaluate how treatment with Kinetic Oscillation Stimulation (KOS) in the nasal cavity in patients with non-allergic rhinitis can be optimized to minimize any patient reported discomfort during treatment procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent (>12w) symptoms of idiopathic rhinitis dominated by nasal congestion (± secretion) for an average of at least 1 h per day for at least 5 days during a period of 14 days
* Having nasal congestion as major symptom, and a nasal congestion score of at least 2 (scale 0-3)
* Male or female 18 - 65 years
* Judged by the Investigator as suitable for participation in the study without safety concerns based on medical history and physical examination
* Willing and able to provide written informed consent prior to participation in the clinical investigation
* Willing and able to comply with all study related procedure

Exclusion Criteria:

* Patients with Allergic rhinitis, demonstrated by either positive skin prick test, phadiatop or RAST(radioallergosorbent test)
* Ongoing respiratory tract infection including nasal cavity at inclusion (treatment visit 1)
* Systemic steroid treatment less than 4 weeks before the inclusion in the study
* Patients with a history of nasal surgery like: septoplasty, cosmetic surgery, conchal surgery or any other nasal surgery except closed reposition for nasal fracture
* History of frequent nose bleeds or a condition that increases the risk of excessive bleeding
* Pronounced anterior septal deviation or other significant nasal pathology at endoscopic examination
* Current malignancy of any kind
* Known allergy to polyvinylchloride or medicinal liquid paraffin
* Any disease, condition (medical or surgical) which, in the opinion of the investigator, might compromise the study results, or would place the subject at increased risk
* Any implant with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, defibrillator, vagal neurostimulator, deep brain stimulation, spinal stimulator, bone growth stimulator, or cochlear implant or any other implant in the head-, and neck region
* Previous treated with radiation on the face, head or neck regions
* Female patients who are pregnant or nursing, or become pregnant at any time from first visit at ENT(Ear, Nose and Throat) - clinic until treatment day (second visit)
* Female patients: unwilling to use adequate contraceptive between first and last visit
* Received study drug in a clinical trial for an investigational drug within the previous 30 days, or 5 half-lives, whichever is longer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pain score on the Visual Analogue Scale | Five seconds after placement of catheter in nasal cavity
  To evaluate whether patient´s self-administration of catheter into nasal cavity is associated with a different degree of patient-reported pain on Visual Analogue Scales (VAS) compared to when administered by a health professional.

SECONDARY OUTCOMES:
Sino-Nasal Outcome Test-22 (SNOT-22) questionnaire | Baseline, day 14
  To evaluate if treatment effect (assessed 15 minutes before treatment and 14 days after treatment) by SNOT-22 is different between treatment groups.

OTHER OUTCOMES:
Peak Nasal Inspiratory Flow (PNIF) | Baseline, day 14
  To evaluate if treatment effect (assessed 15 minutes before treatment and 14 days after treatment) by PNIF is different between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Finn Jorgensen, M.D., Ph.D., Principal Investigator — Halmstad County Hospital
Locations (1):
- Ear, Nose and Throat Dept, Halmstad County Hospital, Halmstad, Sweden